CLINICAL TRIAL: NCT05772299
Title: Treatment of Peri-implant Mucositis Using an Er:Yag Laser or an Ultrasonic Device. A Randomized Clinical Trial
Brief Title: Treatment of Inflammation Around Implants With a Laser or an Ultrasonic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Viveca Wallin Bengtsson, Principle investigator, Kristianstad University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-I mucositis
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Peri-implant Mucositis
Keywords: Clinical study; Bleeding on probing; Pus; Er:Yag laser; Ultrasonic device
MeSH Terms: conditions — Suppuration | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: Test group: will be treated using the Er:Yag laser device (AdvErL EVO, Morita Corporation, Japan). The tip is placed in the pocket mesially, lingually, distally and buccally.
  Control group: will be treated using an ultrasonic device with PEEK coated tips (EMS, Switzerland). The tip is placed in the pocket mesially, lingually, distally and buccally.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor, in this case the dental hygienist performing the registrations/measurement, is blinded during the whole study
  The principal investigator, in this case the periodontologist performing all the treatments, and is therefore not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er:Yag laser treatment (Experimental): The experimental (test) group will receive the following treatment:
  The submucosal debridement will be performed with an Er:Yag laser (AdvErL EVO, Morita Corporation, Japan). The P-400 tip is placed into the peri-implant mucositis pockets mesially, lingually, distally and buccally while rinsing water. Careful attempts are to cover the full circumference of the implant.
  Interventions: Radiation: Er:Yag laser
- Ultrasonic device treatment (Active Comparator): The active comparator (control) group will receive the following treatment:
  The submucosal debridement will be performed by a piezoelectric ultrasonic device with a PEEK coated tip (EMS, Switzerland). The tip is placed into the peri-implant mucositis pockets mesially, lingually, distally and buccally while rinsing water. Careful attempts are to cover the full circumference of the implant.
  Interventions: Device: EMS ultrasound

INTERVENTIONS:
Radiation: Er:Yag laser — Submucosal debridement is performed with Er:Yag laser using a P-400 tip under rinsing water.
  Arms: Er:Yag laser treatment
Device: EMS ultrasound — Submucosal debridement is performed with piezoelectric ultrasound (EMS) with a PEEK (plastic coated) tip under rinsing water.
  Arms: Ultrasonic device treatment

SUMMARY:
The goal of the clinical trial is to compare laser therapy with ultrasonic therapy in patients with inflammation in the tissue surrounding single implants (peri-implant mucositis). The outcomes are bleeding on probing (BOP), pocket depth, suppuration, recession of the peri-implant mucosal margin, the treatment time and changes in bone levels before and after treatment in the test, and control group respectively. The quality of life will be measured from a standardized protocol.

The hypothesis is that treatment with laser therapy in patients with peri-implant mucositis will show less inflammation with less bleeding and a better pocket closure compared to the treatment with the ultrasound.

DETAILED DESCRIPTION:
Data from the clinical treatment will be registered in medical records. In parallel, clinical data will be documented in a study protocol and saved in a safe together with a code list in accordance with a standard operation procedure at the clinic.The protocol with the specific treatment procedure (test or control) will not be opened until the study is completed and only by authorized persons with access to the data in the study such as, the principal investigator and the statisticians.

Variables used in the study originates from an international world workshop on the classification of periodontal and peri-implant diseases and conditions in 2018. In accordance with the working group a diagnosis of peri-implant mucositis should include bleeding on probing and or pus and no bone loss (X-ray). In this study the primary outcomes are bleeding on probing (BOP) and or pus and pocket depth,

The aim is to assess the clinical outcome over 6 months following treatment with non-surgical debridement using an Er:Yag laser device (AdvErL EVO, Morita corporation, Japan) (Test group) or with the use of mechanical therapy using an ultrasonic device with a specially designed tip (EMS, Switzerland) (Control group). An active comparator (Control group) was compared to an experimental arm (Test group).

Patients will therefore be randomized into a test or control group. Inclusion criteria will follow a full mouth routine periodontal examination, including analysis of available radiographs.

All measurements will be performed by a dental hygienist who is blinded for the specific treatment test or control. A periodontist will perform all the treatments and is therefore not blinded. Upon the final appointment the specific arm of treatment will be registered by the periodontist in the patient journal.

All patients will be given oral and written information about the study and sign a written informed consent. The patients will be informed that they could drop off whenever they want without any explanations. The ethical board approved the study.

The test group will be treated using the Er:Yag laser device.The control group will be treated using an ultrasonic device with peek coated tips (EMS, Switzerland). Following treatment all patients, independent of group, will be instructed in proper home care using a toothbrush and interproximal aids as needed.

Study design:

* Baseline: Clinical registrations and treatment
* 1 month: Clinical registrations
* 3 months: Clinical registrations and treatment
* 6 months: Clinical registrations and treatment

In addition, the instrument Oral Health Impact Profile (OHIP) will be used as a measurement of quality of life.

Adverse events will be evaluated at each visit. If a patient should require any treatment during the study the necessary treatment will be provided and according to the standard of care. If adverse events related to the treatment they will be recorded. The investigation will be performed according to the principles of the Declaration of Helsinki on experimentation involving human subjects.

Participant not fulfilling the study will be reported in the patient journal as not completed and statistically noted as missing data.

From the statistical power analysis 38 individuals were minimum to reach a clinically significant difference. The power analysis was based on: if bleeding on probing (BOP) is reduced with 30% ± 10 in the test group and with a 30% decrease in the control group is to be detected at alpha =0.05 and a power of beta= 0.2. Hence it is foreseen to incorporate 45 subjects in the study if some of the individuals will not fulfil the study.

The IBM SPSS version 28.0 statistical software package (SPSS Inc., Armonk, NY, USA) for personal computer will be used in the statistical analyses.

Statistics will be calculated as means with standard deviation (SD). Independent t-tests (equal variance not assumed) paired t-test and one-way ANOVA test will be used to compare inter and intra-group differences. Non-parametric chi-square test will be used for categorical variables. Statistical significance will be set with 80 percent at p < 0.05. Non visits will be recorded as missing data in the statistics.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 1 peri-implant site with probing depth ≥ 4 mm combined with bleeding and or pus on probing
* bone loss ≤ 2 mm measured from the implant shoulder (as a consequence of remodelling during the healing process)

Exclusion Criteria:

* Subjects with uncontrolled diabetes HbA1c >6.5
* Subjects requiring prophylactic antibiotics
* Subjects taking prednisolone
* Subjects taking medications known to have effects on gingival overgrowth

Ages: 23 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | Baseline
  millimeter
Bleeding on probing (BOP) | 1 month
  millimeter
Bleeding on probing (BOP) | 3 months
  millimeter
Bleeding on probing (BOP) | 6 months
  millimeter
Probing pocket depth (PPD) | Baseline
  millimeter
Probing pocket depth (PPD) | 1 month
  millimeter
Probing pocket depth (PPD) | 3 months
  millimeter
Probing pocket depth (PPD) | 6 months
  millimeter
Pus | Baseline
  Presence or abscence
Pus | 1 month
  Presence or abscence
Pus | 3 months
  Presence or abscence
Pus | 6 months
  Presence or abscence

SECONDARY OUTCOMES:
Recession of the peri-implant mucosal margin | Baseline
  millimeter
Recession of the peri-implant mucosal margin | 6 months
  millimeter
Bone level (peri-apical radiographs) | Baseline
  millimeter on Xray
Bone level (peri-apical radiographs) | 6 months
  millimeter on Xray
Implant loss | Baseline
  Prevalence
Implant loss | 1 month
  Prevalence
Implant loss | 3 months
  Prevalence
Implant loss | 6 months
  Prevalence
Treatment time | Baseline
  minutes
Treatment time | 3 months
  minutes
Treatment time | 6 months
  minutes
Quality of life (QoL) | Baseline
  Questionnaire "Oral Health Impact Proflie" (OHIP-14) on a 5 -point Likert scale 0=never (best) ; 5=very often (worst)
Quality of life (QoL) | 6 months
  Questionnaire "Oral Health Impact Profile" (OHIP-14) on a 5 -point Likert scale 0=never (best) ; 5=very often (worst)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Renvert, Prof, Principal Investigator — Kristianstad University
Locations (1):
- University of Kristianstad, Kristianstad, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aoki A, Sasaki KM, Watanabe H, Ishikawa I. Lasers in nonsurgical periodontal therapy. Periodontol 2000. 2004;36:59-97. doi: 10.1111/j.1600-0757.2004.03679.x. No abstract available. PMID 15330944
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Lin GH, Suarez Lopez Del Amo F, Wang HL. Laser therapy for treatment of peri-implant mucositis and peri-implantitis: An American Academy of Periodontology best evidence review. J Periodontol. 2018 Jul;89(7):766-782. doi: 10.1902/jop.2017.160483. PMID 30133748
- [Background] Renvert S, Lessem J, Dahlen G, Lindahl C, Svensson M. Topical minocycline microspheres versus topical chlorhexidine gel as an adjunct to mechanical debridement of incipient peri-implant infections: a randomized clinical trial. J Clin Periodontol. 2006 May;33(5):362-9. doi: 10.1111/j.1600-051X.2006.00919.x. PMID 16634959
- [Background] Renvert S, Persson GR, Pirih FQ, Camargo PM. Peri-implant health, peri-implant mucositis, and peri-implantitis: Case definitions and diagnostic considerations. J Periodontol. 2018 Jun;89 Suppl 1:S304-S312. doi: 10.1002/JPER.17-0588. PMID 29926953
- [Background] Takasaki AA, Aoki A, Mizutani K, Kikuchi S, Oda S, Ishikawa I. Er:YAG laser therapy for peri-implant infection: a histological study. Lasers Med Sci. 2007 Sep;22(3):143-57. doi: 10.1007/s10103-006-0430-x. Epub 2007 Jan 12. PMID 17219255
- [Derived] Bengtsson VW, Aoki A, Mizutani K, Lindahl C, Renvert S. Treatment of peri-implant mucositis using an Er:YAG laser or an ultrasonic device: a randomized, controlled clinical trial. Int J Implant Dent. 2025 Jan 24;11(1):6. doi: 10.1186/s40729-025-00591-0. PMID 39853624

DOCUMENTS (3):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT05772299/Prot_003.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT05772299/SAP_004.pdf
  • Informed Consent Form (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT05772299/ICF_005.pdf